CLINICAL TRIAL: NCT02781181
Title: Carotid Artery Stenting Without Embolic Protection: A Randomized Multicenter Trial (the CASWEP Trial)
Brief Title: Carotid Artery Stenting Without Protection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AcibademU
Record Dates: First submitted 2016-05-16; First posted 2016-05-24 (Estimated); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Carotid Arteries
Keywords: Stenting; Protection device; EPD usage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAS with CPD (Other): CAS performed under neuroprotection
  Interventions: Device: CAS with CPD
- CAS without CPD (Active Comparator): CAS without neuroprotection
  Interventions: Other: CAS without CPD

INTERVENTIONS:
Device: CAS with CPD — using a neuroprotection device
  Arms: CAS with CPD
Other: CAS without CPD — No Neuroprotection
  Arms: CAS without CPD

SUMMARY:
A recent randomized Carotid artery stenting (CAS) trial in which carotid protection device (CPD)s were used to demonstrate equivalence with carotid endarterectomy (CEA) by achieving noninferiority regarding periprocedural risk. However, the clinical efficacy and safety of CPDs are still a matter of controversy. It has been argued that the limited reduction provided by CPDs may be due to the devices themselves. Probably, they serve as sources for emboli during the procedure or removal technique. In general, 30- day adverse outcome for CAS with the use of CPDs seems not to be different from the outcome without CPDs.

Thus, the main goal in this study is to test the hypothesis that CAS without CPD usage is as safe as in those patients who undergo CAS with CPD neuroprotection.

DETAILED DESCRIPTION:
The Carotid Artery Stenting without Embolic Protection (CASWEP) trial is designed in a prospective, randomized, multi-center fashion to determine if CAS without CPD is feasible and safe in patients with symptomatic or asymptomatic severe carotid stenosis.

Study participants After the exclusion criterias were applied 279 patients were divided as 139 patients in the CAS with CPD arm and 140 patients in the CAS without CPD arm. Our study population includes patients with severe carotid artery stenosis referred to the 3 study center hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients with ≥ 50% ipsilateral carotid stenosis by angiography, ≥70% by duplex ultrasound, or ≥70% by Computerized tomography (CT) angiography or Magnetic Resonance (MR) angiography if the stenosis on ultrasonography was 50% to 69%.
* Asymptomatic patients with ≥60% stenosis by angiography, ≥70% by ultrasound, or ≥80% by CT angiography or MR angiography if the stenosis on ultrasonography was 50% to 69%.

Exclusion Criteria:

* Total occlusion,
* Visible thrombus at the lesion site
* Bleeding diathesis
* Cerebral vascular malformation,
* Degenerative cerebral diseases
* Cerebral tumors
* Illness impeding informed consent
* Life expectancy<2 years
* Previous CEA.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2016-05; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
The number of patients experiencing new ischemic brain lesions on diffusion-weighted magnetic resonance imaging (DWMRI), transient ischemic attack (TIA), Stroke and death events. | through hospital admission, an average of 2 days
  peri-procedural in hospital outcome

CONTACTS AND LOCATIONS:
Overall Officials: SEVKET GORGULU, MD, Study Director — Acibadem University
Locations (6):
- Turkey (Türkiye) (6):
  - Adapazari Education and Research Hospital, Adapazarı
  - Adiyaman University, Adıyaman
  - Acibadem University, Istanbul
  - Koşuyolu Training and Research Hospital, Istanbul
  - Marmara University, Istanbul
  - Mehmet Akif Ersoy Education and Training Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gorgulu S, Sahin M, Norgaz NT, Pala S, Sari M, Yalcin AA, Sipahi I. Carotid artery stenting without embolic protection: A randomized multicenter trial (the CASWEP trial). Interv Neuroradiol. 2023 Aug;29(4):419-425. doi: 10.1177/15910199221094388. Epub 2022 Apr 26. PMID 35469509